CLINICAL TRIAL: NCT01548820
Title: Pretreatment and On-treatment Indicators of Virologic Breakthrough in Chronic HBV Egyptian Patients Receiving Lamivudine Therapy
Brief Title: Resistance to Lamivudine in HBV Egyptian Patients
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Iman Fawzy Montasser, Lecturer of tropical medicine , Ain Shams university, Ain Shams University
Other Study IDs: HBV resistance
Record Dates: First submitted 2012-03-06; First posted 2012-03-08 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Hepatitis B Virus Treatment
Keywords: Hepatitis B virus; Lamivudine; Resistance to treatment
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood samples +/- tissue biopsy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chronic HBV Egyptian patients: chronic HBV patients receiving Lamivudine therapy in hepatology clinic in the National Hepatology & Tropical Medicine Research Institute in Egypt.

SUMMARY:
On treatment parameters for Lamivudine resistance in HBV treated Egyptian patients

DETAILED DESCRIPTION:
Primarily: To study the correlations between the following parameters in adult Egyptian patients with chronic viral hepatitis B before treatment:

* ALT.
* HBeAg.
* HBV-DNA by quantitative PCR.
* Biopsy (if possible). Secondarily: After receiving lamivudine therapy we will identify the impact of these parameters on viral breakthrough at 1 year of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >18 years old
* Egyptian nationality
* Positive serology for HBsAg for more than 6 months
* Positive HBV viremia (above 2000IU/ml).
* Lamivudine monotherapy

Exclusion Criteria:

* Anti-HBcIgM seropositivity
* Positive serology for HCV
* Positive serology for HDV
* Patients complicated with HCC

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic HBV patients receiving Lamivudine therapy in hepatology clinic in the National Hepatology & Tropical Medicine Research Institute in Egypt in the period from 2007- 2011.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2010-06; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Resistance to Lamivudine Therapy | 1 year
  Prevelance of Lamivudine resistance among HBV Egyptian cases pretreatment and on treatment parameters for Lamivudine therapy resistance

CONTACTS AND LOCATIONS:
Locations (1):
- Tropical medicine department, Cairo, Egypt